CLINICAL TRIAL: NCT04452318
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled Study Assessing the Efficacy and Safety of Anti-Spike SARS-CoV-2 Monoclonal Antibodies in Preventing SARS-CoV-2 Infection in Household Contacts of Individuals Infected With SARS-CoV-2
Brief Title: COVID-19 Study Assessing the Efficacy and Safety of Anti-Spike SARS CoV-2 Monoclonal Antibodies for Prevention of SARS CoV-2 Infection Asymptomatic in Healthy Adults and Adolescents Who Are Household Contacts to an Individual With a Positive SARS-CoV-2 RT-PCR Assay
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R10933-10987-COV-2069; 2020-003654-71 (EudraCT Number)
Record Dates: First submitted 2020-06-26; First posted 2020-06-30 (Actual); Results first posted 2023-05-15 (Actual); Last update posted 2023-05-15 (Actual); Status verified 2023-04

CONDITIONS: Healthy Participants
Keywords: Asymptomatic; Individuals at risk of exposure to SARS-CoV-2; Household Contacts of a Person Infected with SARS-CoV-2
MeSH Terms: interventions — casirivimab; imdevimab; casirivimab and imdevimab drug combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- REGN10933 + REGN10987 (Experimental)
  Interventions: Drug: REGN10933 + REGN10987
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: REGN10933 + REGN10987 — Subcutaneous (SC) or Intramuscular (IM) injections
  Other Names: REGN-COV2; Casirivimab; Imdevimab; REGEN-COV™
  Arms: REGN10933 + REGN10987
Drug: Placebo — SC or IM injections
  Arms: Placebo

SUMMARY:
Primary Objectives:

Cohort A:

• To evaluate the efficacy of REGN10933+REGN10987 compared to placebo in preventing symptomatic SARS-CoV-2 infection (broad-term) confirmed by RT-qPCR

Cohort A and Cohort A1:

• To evaluate the safety and tolerability of REGN10933+REGN10987 following subcutaneous (SC) administration compared to placebo

Cohort B • To evaluate the efficacy of REGN10933+REGN10987 compared to placebo in preventing COVID-19 symptoms (broad-term)

Cohort B and Cohort B1

• To evaluate the safety and tolerability of REGN10933+REGN10987 following SC administration compared to placebo

DETAILED DESCRIPTION:
Cohort A: adult and adolescent subjects (≥12 years) who are SARS -CoV-2 RT-qPCR negative at baseline

Cohort A1: pediatric subjects (<12 years) who are SARS-CoV-2 RT--qPCR negative at baseline

Cohort B: adult and adolescent subjects (≥12 years) who are SARS -CoV-2 RT-qPCR positive at baseline

Cohort B1: pediatric subjects (<12 years) who are SARS-CoV-2 RT--qPCR positive at baseline

ELIGIBILITY:
Key Inclusion Criteria:

1. Adult subjects 18 years of age (irrespective of weight) and above at the signing of informed consent or adolescent participants ≥12 to <18 years of age, or pediatric participants <12 years of age at the signing of the assent (parent/guardian sign the informed consent)
2. Asymptomatic household contact with exposure to an individual with a diagnosis of SARS-CoV-2 infection (index case). To be included in the study, participants must be randomized within 96 hours of collection of the index cases' positive SARS-COV-2 diagnostic test sample
3. Participant anticipates living in the same household with the index case until study day 29
4. Is judged by the investigator to be in good health based on medical history and physical examination at screening/baseline, including participants who are healthy or have a chronic, stable medical condition
5. Willing and able to comply with study visits and study-related procedures/assessments.
6. Provide informed consent signed by study participant or legally acceptable representative.

Key Exclusion Criteria:

1. History of prior positive SARS-CoV-2 RT-PCR test or positive SARS-CoV-2 serology test at any time before the screening
2. Participant has lived with individuals who have had previous SARS-CoV-2 infection or currently lives with individuals who have SARS-CoV-2 infection, with the exception of the index case(s), the first individual(s) known to be infected in the household
3. Active respiratory or non-respiratory symptoms consistent with COVID-19
4. History of respiratory illness with sign/symptoms of SARS-CoV-2 infection, in the opinion of the investigator, within the prior 6 months to screening
5. Nursing home resident
6. Any physical examination findings, and/or history of any illness, concomitant medications or recent live vaccines that, in the opinion of the study investigator, might confound the results of the study or pose an additional risk to the participant by their participation in the study

Note: Other protocol-defined Inclusion/ Exclusion criteria apply

Min Age: 1 Day | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 3303 (Actual)
Dates: Start 2020-07-13 (Actual); Primary Completion 2021-10-04 (Actual); Study Completion 2021-10-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (104):
- United States (102):
  - Regeneron Study Site, Mesa, Arizona
  - Regeneron Study Site, Tucson, Arizona
  - Regeneron Study Site, La Mesa, California
  - Regeneron Study Site, La Palma, California
  - Regeneron Study Site, Long Beach, California
  - Regeneron Study Site, Los Angeles, California
  - Regeneron Study Site, Montclair, California
  - Regeneron Study Site, Northridge, California
  - Regeneron Study Site, Oxnard, California
  - Regeneron Study Site, Sacramento, California
  - Regeneron Study Site, San Diego, California
  - Regeneron Study Site, San Francisco, California
  - Regeneron Study Site, Stanford, California
  - Regeneron Study Site, Torrance, California
  - Regeneron Study Site, Aurora, Colorado
  - Regeneron Study Site, Colorado Springs, Colorado
  - Regeneron Study Site, Washington D.C., District of Columbia
  - Regeneron Study Site, Boca Raton, Florida
  - Regeneron Study Site, Clearwater, Florida
  - Regeneron Study Site, DeLand, Florida
  - Regeneron Study Site, Ft. Pierce, Florida
  - Regeneron Study Site, Hialeah, Florida
  - Regeneron Study Site, Jacksonville, Florida
  - Regeneron Study Site, Lakeland, Florida
  - Regeneron Study Site, Loxahatchee Groves, Florida
  - Regeneron Study Site, Maitland, Florida
  - Regeneron Study Site, Miami, Florida
  - Regeneron Study Site, Orlando, Florida
  - Regeneron Study Site, Sarasota, Florida
  - Regeneron Study Site, Tampa, Florida
  - Regeneron Study Site, West Palm Beach, Florida
  - Regeneron Study Site, Winter Park, Florida
  - Regeneron Study Site, Atlanta, Georgia
  - Regeneron Study Site, Columbus, Georgia
  - Regeneron Study Site, Decatur, Georgia
  - Regeneron Study Site, Eatonton, Georgia
  - Regeneron Study Site, Marietta, Georgia
  - Regeneron Study Site, Sandy Springs, Georgia
  - Regeneron Study Site, Chicago, Illinois
  - Regeneron Study Site 2, Chicago, Illinois
  - Regeneron Study Site 3, Chicago, Illinois
  - Regeneron Study Site 1, Downers Grove, Illinois
  - Regeneron Study Site 2, Downers Grove, Illinois
  - Regeneron Study Site, Ames, Iowa
  - Regeneron Study Site, Lake Charles, Louisiana
  - Regeneron Study Site, Marrero, Louisiana
  - Regeneron Study Site, Metairie, Louisiana
  - Regeneron Study Site, New Orleans, Louisiana
  - Regeneron Study Site, Baltimore, Maryland
  - Regeneron Study Site, Boston, Massachusetts
  - Regeneron Study Site, Detroit, Michigan
  - Regeneron Study Site, Royal Oak, Michigan
  - Regeneron Study Site, Minneapolis, Minnesota
  - Regeneron Study Site, Gulfport, Mississippi
  - Regeneron Study Site, Jackson, Mississippi
  - Regeneron Study Site, Hazelwood, Missouri
  - Regeneron Study Site, St Louis, Missouri
  - Regeneron Study Site, Las Vegas, Nevada
  - Regeneron Study Site, Morristown, New Jersey
  - Regeneron Study Site, Newark, New Jersey
  - Regeneron Study Site, Summit, New Jersey
  - Regeneron Study Site, Teaneck, New Jersey
  - Regeneron Study Site, Buffalo, New York
  - Regeneron Study Site, New York, New York
  - Regeneron Study Site 1, The Bronx, New York
  - Regeneron Study Site 2, The Bronx, New York
  - Regeneron Study Site, The Bronx, New York
  - Regeneron Study Site, Chapel Hill, North Carolina
  - Regeneron Study Site, Charlotte, North Carolina
  - Regeneron Study Site, Fayetteville, North Carolina
  - Regeneron Study Site, Raleigh, North Carolina
  - Regeneron Study Site, Wilmington, North Carolina
  - Regeneron Study Site, Winston-Salem, North Carolina
  - Regeneron Study Site, Cincinnati, Ohio
  - Regeneron Study Site, Columbus, Ohio
  - Regeneron Study Site, Dayton, Ohio
  - Regeneron Study Site, Danville, Pennsylvania
  - Regeneron Study Site, Philadelphia, Pennsylvania
  - Regeneron Study Site, Wilkes-Barre, Pennsylvania
  - Regeneron Study Site, Providence, Rhode Island
  - Regeneron Study Site, Charleston, South Carolina
  - Regeneron Study Site, Clinton, South Carolina
  - Regeneron Study Site, Gaffney, South Carolina
  - Regeneron Study Site, Sioux Falls, South Dakota
  - Regeneron Study Site, Chattanooga, Tennessee
  - Regeneron Study Site, Knoxville, Tennessee
  - Regeneron Study Site, Memphis, Tennessee
  - Regeneron Study Site, Nashville, Tennessee
  - Regeneron Study Site, Bellaire, Texas
  - Regeneron Study Site, Corpus Christi, Texas
  - Regeneron Study Site, Dallas, Texas
  - Regeneron Study Site, Houston, Texas
  - Regeneron Study Site, Pearland, Texas
  - Regeneron Study Site, Red Oak, Texas
  - Regeneron Study Site, San Antonio, Texas
  - Regeneron Study Site, Tyler, Texas
  - Regeneron Study Site, Charlottesville, Virginia
  - Regeneron Study Site, Richmond, Virginia
  - Regeneron Study Site, Everett, Washington
  - Regeneron Study Site, Seattle, Washington
  - Regeneron Study Site, Yakima, Washington
  - Regeneron Study Site, Madison, Wisconsin
- Regeneron Study Site, Chisinau, Moldova
- Regeneron Study Site, Bucharest, Romania

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Individual anonymized participant data will be considered for sharing once the indication has been approved by a regulatory body, if there is legal authority to share the data and there is not a reasonable likelihood of participant re-identification.
Access Criteria: Qualified researchers may request access to anonymized patient level data or aggregate study data when Regeneron has received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency [EMA], Pharmaceuticals and Medical Devices Agency [PMDA], etc) for the product and indication, has the legal authority to share the data, and has made the study results publicly available (eg, scientific publication, scientific conference, clinical trial registry).
URL: https://vivli.org/

REFERENCES:
- [Derived] Follmann D, O'Brien MP, Fintzi J, Fay MP, Montefiori D, Mateja A, Herman GA, Hooper AT, Turner KC, Chan KC, Forleo-Neto E, Isa F, Baden LR, El Sahly HM, Janes H, Doria-Rose N, Miller J, Zhou H, Dang W, Benkeser D, Fong Y, Gilbert PB, Marovich M, Cohen MS. Examining protective effects of SARS-CoV-2 neutralizing antibodies after vaccination or monoclonal antibody administration. Nat Commun. 2023 Jun 17;14(1):3605. doi: 10.1038/s41467-023-39292-w. PMID 37330602
- [Derived] Herman GA, O'Brien MP, Forleo-Neto E, Sarkar N, Isa F, Hou P, Chan KC, Bar KJ, Barnabas RV, Barouch DH, Cohen MS, Hurt CB, Burwen DR, Marovich MA, Musser BJ, Davis JD, Turner KC, Mahmood A, Hooper AT, Hamilton JD, Parrino J, Subramaniam D, Baum A, Kyratsous CA, DiCioccio AT, Stahl N, Braunstein N, Yancopoulos GD, Weinreich DM; COVID-19 Phase 3 Prevention Trial Team. Efficacy and safety of a single dose of casirivimab and imdevimab for the prevention of COVID-19 over an 8-month period: a randomised, double-blind, placebo-controlled trial. Lancet Infect Dis. 2022 Oct;22(10):1444-1454. doi: 10.1016/S1473-3099(22)00416-9. Epub 2022 Jul 5. PMID 35803290
- [Derived] Hirsch C, Park YS, Piechotta V, Chai KL, Estcourt LJ, Monsef I, Salomon S, Wood EM, So-Osman C, McQuilten Z, Spinner CD, Malin JJ, Stegemann M, Skoetz N, Kreuzberger N. SARS-CoV-2-neutralising monoclonal antibodies to prevent COVID-19. Cochrane Database Syst Rev. 2022 Jun 17;6(6):CD014945. doi: 10.1002/14651858.CD014945.pub2. PMID 35713300
- [Derived] O'Brien MP, Forleo-Neto E, Sarkar N, Isa F, Hou P, Chan KC, Musser BJ, Bar KJ, Barnabas RV, Barouch DH, Cohen MS, Hurt CB, Burwen DR, Marovich MA, Brown ER, Heirman I, Davis JD, Turner KC, Ramesh D, Mahmood A, Hooper AT, Hamilton JD, Kim Y, Purcell LA, Baum A, Kyratsous CA, Krainson J, Perez-Perez R, Mohseni R, Kowal B, DiCioccio AT, Geba GP, Stahl N, Lipsich L, Braunstein N, Herman G, Yancopoulos GD, Weinreich DM; COVID-19 Phase 3 Prevention Trial Team. Effect of Subcutaneous Casirivimab and Imdevimab Antibody Combination vs Placebo on Development of Symptomatic COVID-19 in Early Asymptomatic SARS-CoV-2 Infection: A Randomized Clinical Trial. JAMA. 2022 Feb 1;327(5):432-441. doi: 10.1001/jama.2021.24939. PMID 35029629
- [Derived] Kreuzberger N, Hirsch C, Chai KL, Tomlinson E, Khosravi Z, Popp M, Neidhardt M, Piechotta V, Salomon S, Valk SJ, Monsef I, Schmaderer C, Wood EM, So-Osman C, Roberts DJ, McQuilten Z, Estcourt LJ, Skoetz N. SARS-CoV-2-neutralising monoclonal antibodies for treatment of COVID-19. Cochrane Database Syst Rev. 2021 Sep 2;9(9):CD013825. doi: 10.1002/14651858.CD013825.pub2. PMID 34473343
- [Derived] O'Brien MP, Forleo-Neto E, Musser BJ, Isa F, Chan KC, Sarkar N, Bar KJ, Barnabas RV, Barouch DH, Cohen MS, Hurt CB, Burwen DR, Marovich MA, Hou P, Heirman I, Davis JD, Turner KC, Ramesh D, Mahmood A, Hooper AT, Hamilton JD, Kim Y, Purcell LA, Baum A, Kyratsous CA, Krainson J, Perez-Perez R, Mohseni R, Kowal B, DiCioccio AT, Stahl N, Lipsich L, Braunstein N, Herman G, Yancopoulos GD, Weinreich DM; Covid-19 Phase 3 Prevention Trial Team. Subcutaneous REGEN-COV Antibody Combination to Prevent Covid-19. N Engl J Med. 2021 Sep 23;385(13):1184-1195. doi: 10.1056/NEJMoa2109682. Epub 2021 Aug 4. PMID 34347950
- [Derived] O'Brien MP, Forleo-Neto E, Musser BJ, Isa F, Chan KC, Sarkar N, Bar KJ, Barnabas RV, Barouch DH, Cohen MS, Hurt CB, Burwen DR, Marovich MA, Hou P, Heirman I, Davis JD, Turner KC, Ramesh D, Mahmood A, Hooper AT, Hamilton JD, Kim Y, Purcell LA, Baum A, Kyratsous CA, Krainson J, Perez-Perez R, Mohseni R, Kowal B, DiCioccio AT, Stahl N, Lipsich L, Braunstein N, Herman G, Yancopoulos GD, Weinreich DM. Subcutaneous REGEN-COV Antibody Combination for Covid-19 Prevention. medRxiv [Preprint]. 2021 Jun 17:2021.06.14.21258567. doi: 10.1101/2021.06.14.21258567. PMID 34159344
- [Derived] O'Brien MP, Forleo-Neto E, Sarkar N, Isa F, Hou P, Chan KC, Musser BJ, Bar KJ, Barnabas RV, Barouch DH, Cohen MS, Hurt CB, Burwen DR, Marovich MA, Brown ER, Heirman I, Davis JD, Turner KC, Ramesh D, Mahmood A, Hooper AT, Hamilton JD, Kim Y, Purcell LA, Baum A, Kyratsous CA, Krainson J, Perez-Perez R, Mohseni R, Kowal B, DiCioccio AT, Stahl N, Lipsich L, Braunstein N, Herman G, Yancopoulos GD, Weinreich DM; COVID-19 Phase 3 Prevention Trial Team. Subcutaneous REGEN-COV Antibody Combination in Early Asymptomatic SARS-CoV-2 Infection: A Randomized Clinical Trial. medRxiv [Preprint]. 2021 Sep 18:2021.06.14.21258569. doi: 10.1101/2021.06.14.21258569. PMID 34159343

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 3375 participants screened, 3298 participants were randomized and 3270 participants were treated. 77 participants were screen failures and 28 participants were randomized but not treated.
Groups:
- Cohort A: Placebo of R10933 + R10987: Cohort A: Placebo of R10933 + R10987 Adult and Adolescent Subjects (≥12years) Who Are SARS-CoV-2 RT-qPCR negative at baseline
- R10933 + R10987: R10933 + R10987 Adult and Adolescent Subjects (≥12years) Who Are SARS-CoV-2 RT-qPCR negative at baseline
- Cohort A1: Placebo of R10933 + R10987: Cohort A1: Placebo of R10933 + R10987 Pediatric Subjects (<12 years) with SARS-CoV-2 RT-qPCR Negative
- Cohort B: Placebo of R10933 + R10987: Cohort B: Placebo of R10933 + R10987 Adult and Adolescent Subjects (≥12years) Who Are SARS-CoV-2 RT-qPCR Positive
- Cohort B: R10933 + R10987: Cohort B: R10933 + R10987 Adult and Adolescent Subjects (≥12years) who Are SARS-CoV-2 RT-qPCR Positive
- Undetermined: Placebo of R10933 + R10987: Undetermined: Placebo of R10933 + R10987 Adult and Adolescent subjects (≥12 years) whose baseline RT-qPCR status was inconclusive or missing
- Undetermined: R10933 + R10987: Undetermined: R10933 + R10987 Adult and Adolescent subjects (≥12 years) whose baseline RT-qPCR status was inconclusive or missing
Period: Overall Study
Arm/Group | Cohort A: Placebo of R10933 + R10987 | R10933 + R10987 | Cohort A1: Placebo of R10933 + R10987 | Cohort B: Placebo of R10933 + R10987 | Cohort B: R10933 + R10987 | Undetermined: Placebo of R10933 + R10987 | Undetermined: R10933 + R10987
Started | 1430 | 1441 | 1 | 173 | 166 | 53 | 34
Randomized and Treated | 1428 | 1439 | 1 | 170 | 165 | 44 | 23
Completed | 1343 | 1368 | 1 | 150 | 157 | 41 | 22
Not Completed | 87 | 73 | 0 | 23 | 9 | 12 | 12
Not completed — Physician Decision | 1 | 2 | 0 | 2 | 0 | 2 | 5
Not completed — Death | 2 | 3 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 38 | 28 | 0 | 3 | 3 | 2 | 1
Not completed — Withdrawal by Subject | 46 | 40 | 0 | 18 | 6 | 8 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A: Placebo of R10933 + R10987 | R10933 + R10987 | Cohort A1: Placebo of R10933 + R10987 | Cohort B: Placebo of R10933 + R10987 | Cohort B: R10933 + R10987 | Undetermined: Placebo of R10933 + R10987 | Undetermined: R10933 + R10987 | Total
Number analyzed (Participants) | 1430 | 1441 | 1 | 173 | 166 | 53 | 34 | 3298
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.4 (15.70) | 42.1 (16.00) | 10.0 (0.0) | 41.8 (18.1) | 39.5 (17.81) | 43.0 (16.73) | 39.0 (15.3) | 42.0 (16.10)
Age, Customized [Count of Participants; unit: Participants]
  In utero | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Preterm newborn infants (gestational age < 37 wks) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Newborns (0-27 days) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Infants and toddlers (28 days-23 months) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Children (2-11 years) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Adolescents (12-17 years) | 47 | 52 | 0 | 20 | 23 | 2 | 1 | 145
  Adults (18-64 years) | 1272 | 1263 | 0 | 130 | 127 | 45 | 30 | 2867
  From 65-84 years | 105 | 125 | 0 | 21 | 15 | 5 | 3 | 274
  85 years and over | 6 | 1 | 0 | 2 | 1 | 1 | 0 | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 738 | 780 | 0 | 97 | 80 | 21 | 20 | 1736
  Male | 692 | 661 | 1 | 76 | 86 | 32 | 14 | 1562
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 707 | 698 | 1 | 66 | 69 | 23 | 9 | 1573
  Not Hispanic or Latino | 711 | 735 | 0 | 105 | 96 | 30 | 25 | 1702
  Unknown or Not Reported | 12 | 8 | 0 | 2 | 1 | 0 | 0 | 23
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 1193 | 1196 | 1 | 149 | 140 | 46 | 29 | 2754
  Black or African American | 161 | 164 | 0 | 11 | 9 | 4 | 1 | 350
  Asian | 37 | 42 | 0 | 8 | 11 | 3 | 2 | 103
  American Indian or Alaska Native | 5 | 4 | 0 | 1 | 1 | 0 | 0 | 11
  Native Hawaiian or Other Pacific Islander | 2 | 3 | 0 | 0 | 0 | 0 | 0 | 5
  Other | 32 | 32 | 0 | 4 | 5 | 0 | 2 | 75

OUTCOME MEASURES:

1. Primary Outcome: Cohort A: Percentage of Participants Who Have a Symptomatic RT-qPCR Confirmed SARS-CoV-2 Infection (Broad-term) During the EAP
Description: Symptomatic SARS-CoV-2 infection (broad-term) is defined as a positive central lab SARS-CoV-2 RT-qPCR result (either NP, nasal or saliva) associated with signs and symptoms with the onset date occurring within 14 days of a positive RT-qPCR during the EAP. Percentage estimated by Logistic Regression.
Time Frame: Up to 1 month
Population: Seronegative modified full analysis set in Cohort A includes randomized subjects aged 12 years and older who are laboratory confirmed negative for SARS-CoV-2 and negative serostatus for SAS-CoV-2 antibodies at baseline
Measure: Number; unit: Percentage of Participants
Groups:
- Cohort A: R10933 + R10987: Cohort A: R10933 + R10987 Adult and Adolescent Subjects (≥12years) Who Are SARS-CoV-2 RT-qPCR negative at baseline
Arm/Group | Cohort A: Placebo of R10933 + R10987 | Cohort A: R10933 + R10987
Number analyzed (Participants) | 752 | 753
Percentage of Participants | 7.8 | 1.4
Statistical Analysis 1: Comparison: Cohort A: Placebo of R10933 + R10987 vs Cohort A: R10933 + R10987; Test type: Superiority; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 0.17, 95% CI 2-sided [0.090 to 0.332]

2. Primary Outcome: Cohort B: Percentage of Participants Who Subsequently Develop Signs and Symptoms (Broad-Term) Within 14 Days of a Positive RT-qPCR at Baseline or During the EAP
Description: The percentage of participants was estimated by using the logistic regression model with fixed categorical effects of treatment group, age group (age in years:>=12 to=50), and region (US vs ex-US).
Time Frame: Up to 14 Days
Population: Estimate of percent of participants meeting the criteria based on fixed categories
Measure: Number; unit: Percentage of Participants
Arm/Group | Cohort B: Placebo of R10933 + R10987 | Cohort B: R10933 + R10987
Number analyzed (Participants) | 104 | 100
Percentage of Participants | 42.5 | 28.4
Statistical Analysis 1: Comparison: Cohort B: Placebo of R10933 + R10987 vs Cohort B: R10933 + R10987; Test type: Superiority; p = 0.0380, Regression, Logistic; Odds Ratio (OR) = 0.54, 95% CI 2-sided [0.298 to 0.966]

3. Primary Outcome: Cohort A and Cohort B: Number of Participants With at Least One Treatment-emergent Adverse Event (TEAEs) and Severity of TEAEs
Time Frame: Up to 8 months
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: Placebo of R10933 + R10987 | Cohort A: R10933 + R10987 | Cohort B: Placebo of R10933 + R10987 | Cohort B: R10933 + R10987
Number analyzed (Participants) | 1428 | 1439 | 170 | 165
Participants
  # of participants with at least one TEAE | 512 | 405 | 88 | 60
  # of participants with at least one Grade 1 TEAE | 384 | 284 | 61 | 51
  # of participants with at least one Grade 2 TEAE | 98 | 95 | 21 | 7
  # of participants with at least one Grade 3 TEAE | 26 | 21 | 6 | 2
  # of participants with at least one Grade 4 TEAE | 2 | 2 | 0 | 0
  # of participants with at least one Grade 5 TEAE | 2 | 3 | 0 | 0

4. Secondary Outcome: Cohort A and Cohort B: Percentage of Participants With High Viral Load in Nasopharyngeal (NP) Swab Samples During the EAP
Description: High viral load (> 4 log 10 copies/ml)
Time Frame: Up to 1 month
Measure: Number; unit: Percentage of Participants
Arm/Group | Cohort A: Placebo of R10933 + R10987 | Cohort A: R10933 + R10987 | Cohort B: Placebo of R10933 + R10987 | Cohort B: R10933 + R10987
Number analyzed (Participants) | 749 | 745 | 101 | 98
Percentage of Participants | 11.3 | 1.6 | 62.6 | 40.5
Statistical Analysis 1: Comparison: Cohort A: Placebo of R10933 + R10987 vs Cohort A: R10933 + R10987; Test type: Superiority; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 0.13, 95% CI 2-sided [0.069 to 0.236]
Statistical Analysis 2: Comparison: Cohort B: Placebo of R10933 + R10987 vs Cohort B: R10933 + R10987; Test type: Superiority; p = 0.0024, Regression, Logistic; Odds Ratio (OR) = 0.41, 95% CI 2-sided [0.228 to 0.728]

5. Secondary Outcome: Cohort A: Number of Weeks of Symptomatic RT-qPCR Confirmed SARS-CoV-2 Infection (Broad Term) During the EAP
Time Frame: Up to 1 month
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | Cohort A: Placebo of R10933 + R10987 | Cohort A: R10933 + R10987
Number analyzed (Participants) | 752 | 753
weeks | 0.25 (1.135) [lower limit 1.135] | 0.02 (0.181) [lower limit 0.181]
Statistical Analysis 1: Comparison: Cohort A: Placebo of R10933 + R10987 vs Cohort A: R10933 + R10987; Test type: Superiority; p < 0.0001, Stratified Wilcoxon Rank Sum Test

6. Secondary Outcome: Cohort A and Cohort B: Number of Weeks of High Viral Load in NP Swab Samples During the EAP
Description: High viral load (> 4 log 10 copies/ml)
Time Frame: Up to 1 month
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | Cohort A: Placebo of R10933 + R10987 | Cohort A: R10933 + R10987 | Cohort B: Placebo of R10933 + R10987 | Cohort B: R10933 + R10987
Number analyzed (Participants) | 749 | 745 | 101 | 98
weeks | 0.18 (0.554) [lower limit 0.554] | 0.02 (0.154) [lower limit 0.154] | 0.81 (0.758) [lower limit 0.758] | 0.49 (0.677) [lower limit 0.677]
Statistical Analysis 1: Comparison: Cohort A: Placebo of R10933 + R10987 vs Cohort A: R10933 + R10987; Test type: Superiority; p < 0.0001, Stratified Wilcoxon Rank Sum Test
Statistical Analysis 2: Comparison: Cohort B: Placebo of R10933 + R10987 vs Cohort B: R10933 + R10987; Test type: Superiority; p = 0.0010, Stratified Wilcoxon Rank Sum Test

7. Secondary Outcome: Cohort A: Number of Weeks of RT-qPCR Confirmed SARS-CoV-2 Infection (Regardless of Symptoms) During the EAP
Time Frame: Up to 1 month
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | Cohort A: Placebo of R10933 + R10987 | Cohort A: R10933 + R10987
Number analyzed (Participants) | 752 | 753
weeks | 0.31 (0.854) [lower limit 0.854] | 0.05 (0.260) [lower limit 0.260]
Statistical Analysis 1: Comparison: Cohort A: Placebo of R10933 + R10987; Test type: Superiority; p < 0.0001, Stratified Wilcoxon Rank Sum Test

8. Secondary Outcome: Cohort A: Percentage of Participants Who Have a RT-qPCR Confirmed SARS-CoV-2 Infection (Regardless of Symptoms) During the EAP
Description: as for outcome 2
Time Frame: Up to 1 month
Population: Estimate of percentage of participants meeting the criteria based on fixed categories
Measure: Number; unit: Percentage of Participants
Arm/Group | Cohort A: Placebo of R10933 + R10987 | Cohort A: R10933 + R10987
Number analyzed (Participants) | 752 | 753
Percentage of Participants | 14.56 | 5.00
Statistical Analysis 1: Comparison: Cohort A: Placebo of R10933 + R10987; Test type: Superiority; p < 0.0001, Multiple Imputation, Logistic Regression; Odds Ratio (OR) = 0.31, 95% CI 2-sided [0.208 to 0.456]

9. Secondary Outcome: Cohort A: Percentage of Participants in Placebo Group With a RT-qPCR Confirmed SARS-CoV-2 Infection During the EAP With an Index Case Participating in Study R10933-10987-COV-2067 (NCT04425629)
Time Frame: Up to 1 month
Measure: Number; unit: Percentage of Participants
Arm/Group | Cohort A: Placebo of R10933 + R10987
Number analyzed (Participants) | 186
Percentage of Participants
  % with index case receiving R10933+R10987 in 2067 | 19.8
  % with index case receiving placebo in 2067 | 19.6
  % with index case treatment in 2067 not available | 10.5

10. Secondary Outcome: Cohort A: Percentage of Participants With a Symptomatic RT-qPCR Confirmed SARS-CoV-2 Infection (CDC Definition) During the EAP
Description: Symptomatic SARS-CoV-2 infection (CDC definition) is defined as a positive central lab SARS-CoV-2 RT-qPCR result (either NP, nasal or saliva) associated with signs and symptoms with the onset date occurring within 14 days of a positive RT-qPCR during the EAP. Percentage estimated by Logistic Regression.
Time Frame: Up to 1 month
Measure: Number; unit: Percentage of participants
Arm/Group | Cohort A: Placebo of R10933 + R10987 | Cohort A: R10933 + R10987
Number analyzed (Participants) | 752 | 753
Percentage of participants | 5.9 | 0.8
Statistical Analysis 1: Comparison: Cohort A: Placebo of R10933 + R10987; Test type: Superiority; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 0.12, 95% CI 2-sided [0.051 to 0.286]

11. Secondary Outcome: Cohort A: Number of Weeks of Symptomatic RT-qPCR-confirmed SARS-CoV-2 Infection (CDC Definition) During the EAP
Time Frame: Up to 1 month
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | Cohort A: Placebo of R10933 + R10987 | Cohort A: R10933 + R10987
Number analyzed (Participants) | 752 | 753
weeks | 0.21 (1.042) [lower limit 1.042] | 0.01 (0.128) [lower limit 0.128]
Statistical Analysis 1: Comparison: Cohort A: Placebo of R10933 + R10987; Test type: Superiority; p < 0.0001, Stratified Wilcoxon Rank Sum Test

12. Secondary Outcome: Cohort A: Percentage of Participants Who Have a Symptomatic RT-qPCR Confirmed SARS-CoV-2 Infection (Strict-term) During the EAP
Description: as for outcome 2
Time Frame: Up to 1 month
Population: Estimate of percentage of participants meeting the criteria based on fixed categories
Measure: Number; unit: Percentage of participants
Arm/Group | Cohort A: Placebo of R10933 + R10987 | Cohort A: R10933 + R10987
Number analyzed (Participants) | 752 | 753
Percentage of participants | 2.8 | 0.2
Statistical Analysis 1: Comparison: Cohort A: Placebo of R10933 + R10987; Test type: Superiority; p = 0.0010, Regression, Logistic; Odds Ratio (OR) = 0.09, 95% CI 2-sided [0.020 to 0.370]

13. Secondary Outcome: Cohort A: Number of Weeks of Symptomatic RT-qPCR Confirmed SARS-CoV-2 Infection (Strict-term) During the EAP
Time Frame: Up to 1 month
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | Cohort A: Placebo of R10933 + R10987 | Cohort A: R10933 + R10987
Number analyzed (Participants) | 752 | 753
weeks | 0.12 (0.843) [lower limit 0.843] | 0.00 (0.084) [lower limit 0.084]
Statistical Analysis 1: Comparison: Cohort A: Placebo of R10933 + R10987; Test type: Superiority; p < 0.0001, Stratified Wilcoxon Rank Sum Test

14. Secondary Outcome: Cohort A: Percentage of Participants Who Have a RT-qPCR Confirmed SARS-CoV-2 Infections at Each Week in the EAP
Time Frame: Week 1, Week 2, Week 3, Week 4
Measure: Number; unit: Percentage of participants
Arm/Group | Cohort A: Placebo of R10933 + R10987 | Cohort A: R10933 + R10987
Number analyzed (Participants) | 752 | 753
Percentage of participants
  Week 1 | 8.9 | 3.1
  Week 2 | 8.5 | 1.1
  Week 3 | 7.7 | 0.7
  Week 4 | 5.6 | 0.7

15. Secondary Outcome: Cohort A: Percentage of Participants Who Have a Symptomatic RT-qPCR Confirmed SARS-CoV-2 Infection (Broad-term) at Each Week in the EAP
Description: as for outcome 2
Time Frame: Week 1, Week 2, Week 3, Week 4
Population: Estimate of percentage of participants meeting the criteria based on fixed categories
Measure: Number; unit: Percentage of participants
Arm/Group | Cohort A: Placebo of R10933 + R10987 | Cohort A: R10933 + R10987
Number analyzed (Participants) | 752 | 753
Percentage of participants
  Week 1 | 5.2 | 1.2
  Week 2 | 4.8 | 0.4
  Week 3 | 3.3 | 0.0
  Week 4 | 2.1 | 0.1

16. Secondary Outcome: Cohort A: Time-weighted Average of Viral Load From the First Positive SARS CoV-2 RT-qPCR in NP Swab Samples (That Has an Onset During the EAP) Until the Third Weekly Visit After the First Positive Test During the EAP
Time Frame: Up to 1 month
Measure: Least Squares Mean (Standard Error); unit: log10 copies/mL
Arm/Group | Cohort A: Placebo of R10933 + R10987 | Cohort A: R10933 + R10987
Number analyzed (Participants) | 107 | 36
log10 copies/mL | 3.065 (0.243) [lower limit 0.243] | 0.942 (0.317) [lower limit 0.317]
Statistical Analysis 1: Comparison: Cohort A: Placebo of R10933 + R10987; Test type: Superiority; p < 0.0001, ANOVA; Difference of LS Means = -2.123, 95% CI 2-sided [-2.707 to -1.539], Standard Error of Mean 0.295

17. Secondary Outcome: Cohort A: Time-weighted Average of Viral Load From the First Positive SARS-CoV-2 RT-qPCR in NP Swab Samples (That Has an Onset During the EAP) Until the Second Weekly Visit After the First Positive Test During the EAP
Time Frame: Up to 1 month
Measure: Least Squares Mean (Standard Error); unit: log10 copies/mL
Arm/Group | Cohort A: Placebo of R10933 + R10987 | Cohort A: R10933 + R10987
Number analyzed (Participants) | 107 | 36
log10 copies/mL | 3.689 (0.281) [lower limit 0.281] | 1.205 (0.368) [lower limit 0.368]
Statistical Analysis 1: Comparison: Cohort A: Placebo of R10933 + R10987; Test type: Superiority; p < 0.0001, ANOVA; Difference of LS Means = -2.483, 95% CI 2-sided [-3.161 to -1.806], Standard Error of Mean 0.342

18. Secondary Outcome: Cohort A: Maximum SARS-CoV-2 RT-qPCR Viral Load in NP Swab Samples Among Individuals With ≥1 RT-qPCR Positive That Has an Onset During the EAP
Time Frame: Up to 1 month
Measure: Least Squares Mean (Standard Error); unit: log10 copies/mL
Arm/Group | Cohort A: Placebo of R10933 + R10987 | Cohort A: R10933 + R10987
Number analyzed (Participants) | 107 | 36
log10 copies/mL | 6.133 (0.301) [lower limit 0.301] | 3.705 (0.402) [lower limit 0.402]
Statistical Analysis 1: Comparison: Cohort A: Placebo of R10933 + R10987; Test type: Superiority; p < 0.0001, ANOVA; Difference of LS Mean = -2.428, 95% CI 2-sided [-3.196 to -1.659], Standard Error of Mean 0.389

19. Secondary Outcome: Cohort A: SARS-CoV-2 RT-qPCR Viral Load in NP Swab Samples Corresponding to the Onset of First Positive RT-qPCR During the EAP
Time Frame: Up to 1 month
Measure: Least Squares Mean (Standard Error); unit: log10 copies/mL
Arm/Group | Cohort A: Placebo of R10933 + R10987 | Cohort A: R10933 + R10987
Number analyzed (Participants) | 107 | 36
log10 copies/mL | 6.141 (0.305) [lower limit 0.305] | 3.700 (0.396) [lower limit 0.396]
Statistical Analysis 1: Comparison: Cohort A: Placebo of R10933 + R10987; Test type: Superiority; p < 0.0001, ANOVA; Difference of LS Mean = -2.441, 95% CI 2-sided [-3.194 to -1.688], Standard Error of Mean 0.381

20. Secondary Outcome: Cohort A: Area Under the Curve (AUC) in Viral Load From the First Positive SARS-CoV-2 RT-qPCR NP Swab Samples Detected During the EAP Until the First Confirmed Negative Test
Time Frame: Up to 1 month
Measure: Mean (Standard Deviation); unit: log10 copies/milliLiter * days
Arm/Group | Cohort A: Placebo of R10933 + R10987 | Cohort A: R10933 + R10987
Number analyzed (Participants) | 81 | 33
log10 copies/milliLiter * days | 65.982 (47.6933) [lower limit 47.6933] | 19.700 (14.8257) [lower limit 14.8257]

21. Secondary Outcome: Cohort A: Total Number of Medically Attended Visits in Emergency Rooms or Urgent Care Centers Related to a RT-qPCR Confirmed SARS-CoV-2 Infection That Has an Onset During the EAP
Description: Medically attended visits referred to hospitalizations, Emergency Room visits, or visits at an Urgent Care center.
Time Frame: Up to 1 month
Measure: Number; unit: medically attended visits
Arm/Group | Cohort A: Placebo of R10933 + R10987 | Cohort A: R10933 + R10987
Number analyzed (Participants) | 752 | 753
medically attended visits | 9 | 0

22. Secondary Outcome: Cohort A: Percentage of Participants With at Least 1 COVID-19-related Hospitalization or Emergency Room Visit Associated With a Positive RT-qPCR During the EAP or All-cause Death
Time Frame: Up to 1 month
Measure: Number; unit: Percentage of Participants
Arm/Group | Cohort A: Placebo of R10933 + R10987 | Cohort A: R10933 + R10987
Number analyzed (Participants) | 752 | 753
Percentage of Participants | 0.5 | 0.0
Statistical Analysis 1: Comparison: Cohort A: Placebo of R10933 + R10987; Testing if there is an association between the observed results and treatment received; Test type: Other; p = 0.0621, Fisher Exact

23. Secondary Outcome: Cohort A: Percentage of Participants Requiring Medically Attended Visits in Emergency Rooms or Urgent Care Centers Related to a RT-qPCR Confirmed SARS CoV-2 Infection That Has an Onset During the EAP
Time Frame: Up to 1 month
Measure: Number; unit: Percentage of participants
Arm/Group | Cohort A: Placebo of R10933 + R10987 | Cohort A: R10933 + R10987
Number analyzed (Participants) | 752 | 753
Percentage of participants | 1.1 | 0.0
Statistical Analysis 1: Comparison: Cohort A: Placebo of R10933 + R10987; Testing if there is an association between the observed results and treatment received'; Test type: Other; p = 0.0038, Fisher Exact

24. Secondary Outcome: Cohort A: Proportion of Participants Hospitalized Related to a RT-qPCR Confirmed SARS-CoV-2 Infection That Has an Onset During the EAP
Description: The proportion of participants hospitalized related to a RT-qPCR confirmed SARS-CoV-2 infection that has an onset during the EAP
Time Frame: Up to 14 Days
Population: Estimate of proportion of participants meeting the criteria based on fixed categories
Measure: Number; unit: Proportion of Participants
Arm/Group | Cohort A: Placebo of R10933 + R10987 | Cohort A: R10933 + R10987
Number analyzed (Participants) | 752 | 753
Proportion of Participants | 0.001 | 0.0

25. Secondary Outcome: Cohort A: Number of Days of Hospital and Intensive Care Unit (ICU) Stay in Participants Hospitalized for a RT-qPCR Confirmed SARS-CoV-2 Infection That Has an Onset During the EAP
Time Frame: Up to Day 29
Population: Only 1 participant in placebo group hospitalized
Measure: Number; unit: Days
Arm/Group | Cohort A: Placebo of R10933 + R10987 | Cohort A: R10933 + R10987
Number analyzed (Participants) | 1 | 0
Days | 11 |

26. Secondary Outcome: Cohort A: Number of Days Missed for Daily Responsibilities Due to a RT-qPCR Confirmed SARS-CoV-2 Infection That Has an Onset During the EAP
Description: Daily responsibilities including work (employed adults) or school (students), daycare or family obligations/responsibilities (childcare or eldercare)
Time Frame: Up to 1 month
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Cohort A: Placebo of R10933 + R10987 | Cohort A: R10933 + R10987
Number analyzed (Participants) | 752 | 753
days | 0.98 (4.659) [lower limit 4.659] | 0.15 (1.276) [lower limit 1.276]
Statistical Analysis 1: Comparison: Cohort A: Placebo of R10933 + R10987; Test type: Superiority; p < 0.0001, Stratified Wilcoxon Rank Sum Test

27. Secondary Outcome: Cohort A: Proportion of Baseline Seropositive Participants (Based on Central Lab Test) With TEAEs and Severity of TEAEs
Time Frame: Up to 8 months
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: Placebo of R10933 + R10987 | Cohort A: R10933 + R10987
Number analyzed (Participants) | 296 | 337
Participants
  with at least one TEAE | 79 | 83
  with at least one serious TEAE | 5 | 6

28. Secondary Outcome: Cohort A and Cohort B: Incidence and Severity of Symptomatic SARS-CoV-2 Infections During the EAP
Time Frame: Up to Day 29
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: Placebo of R10933 + R10987 | Cohort A: R10933 + R10987 | Cohort B: Placebo of R10933 + R10987 | Cohort B: R10933 + R10987
Number analyzed (Participants) | 1428 | 1439 | 170 | 165
Participants
  Total Symptomatic COVID-19 | 81 | 15 | 57 | 35
  Grade 1 Symptomatic COVID-19 | 68 | 11 | 43 | 33
  Grade 2 Symptomatic COVID-19 | 11 | 4 | 12 | 2
  Grade 3 Symptomatic COVID-19 | 2 | 0 | 2 | 0
  Grade 4 Symptomatic COVID-19 | 0 | 0 | 0 | 0
  Grade 5 Symptomatic COVID-19 | 0 | 0 | 0 | 0

29. Secondary Outcome: Cohort A and Cohort B: Incidence and Severity of Symptomatic SARS-CoV-2 Infections During the Follow-Up Period
Time Frame: Day 30 Up to Day 225 (Approximately 8 months)
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: Placebo of R10933 + R10987 | Cohort A: R10933 + R10987 | Cohort B: Placebo of R10933 + R10987 | Cohort B: R10933 + R10987
Number analyzed (Participants) | 1428 | 1439 | 170 | 165
Participants
  Total Symptomatic COVID-19 | 68 | 14 | 1 | 1
  Grade 1 Symptomatic COVID-19 | 50 | 12 | 1 | 1
  Grade 2 Symptomatic COVID-19 | 14 | 2 | 0 | 0
  Grade 3 Symptomatic COVID-19 | 4 | 0 | 0 | 0
  Grade 4 Symptomatic COVID-19 | 0 | 0 | 0 | 0
  Grade 5 Symptomatic COVID-19 | 0 | 0 | 0 | 0

30. Secondary Outcome: Cohort A and Cohort B: Incidence and Severity of Symptomatic SARS-CoV-2 Infections in Seronegative Subjects During the EAP
Time Frame: Up to Day 29
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: Placebo of R10933 + R10987 | Cohort A: R10933 + R10987 | Cohort B: Placebo of R10933 + R10987 | Cohort B: R10933 + R10987
Number analyzed (Participants) | 1067 | 1028 | 114 | 109
Participants
  Total Symptomatic COVID-19 | 74 | 12 | 47 | 32
  Grade 1 Symptomatic COVID-19 | 64 | 9 | 35 | 30
  Grade 2 Symptomatic COVID-19 | 9 | 3 | 10 | 2
  Grade 3 Symptomatic COVID-19 | 1 | 0 | 2 | 0
  Grade 4 Symptomatic COVID-19 | 0 | 0 | 0 | 0
  Grade 5 Symptomatic COVID-19 | 0 | 0 | 0 | 0

31. Secondary Outcome: Cohort A and Cohort B: Incidence and Severity of Symptomatic SARS-CoV-2 Infections in Seronegative Subjects During the Follow-Up Period
Time Frame: Day 30 Up to Day 225 (Approximately 8 months)
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: Placebo of R10933 + R10987 | Cohort A: R10933 + R10987 | Cohort B: Placebo of R10933 + R10987 | Cohort B: R10933 + R10987
Number analyzed (Participants) | 1067 | 1028 | 114 | 109
Participants
  Total Symptomatic COVID-19 | 64 | 10 | 1 | 1
  Grade 1 Symptomatic COVID-19 | 47 | 8 | 1 | 1
  Grade 2 Symptomatic COVID-19 | 14 | 2 | 0 | 0
  Grade 3 Symptomatic COVID-19 | 3 | 0 | 0 | 0
  Grade 4 Symptomatic COVID-19 | 0 | 0 | 0 | 0
  Grade 5 Symptomatic COVID-19 | 0 | 0 | 0 | 0

32. Secondary Outcome: Cohort A and Cohort B: Incidence and Severity of Symptomatic SARS-CoV-2 Infections in Seropositive Subjects During the EAP
Time Frame: Up to Day 29
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: Placebo of R10933 + R10987 | Cohort A: R10933 + R10987 | Cohort B: Placebo of R10933 + R10987 | Cohort B: R10933 + R10987
Number analyzed (Participants) | 296 | 337 | 43 | 48
Participants
  Total Symptomatic COVID-19 | 6 | 3 | 6 | 3
  Grade 1 Symptomatic COVID-19 | 3 | 2 | 5 | 3
  Grade 2 Symptomatic COVID-19 | 2 | 1 | 1 | 0
  Grade 3 Symptomatic COVID-19 | 1 | 0 | 0 | 0
  Grade 4 Symptomatic COVID-19 | 0 | 0 | 0 | 0
  Grade 5 Symptomatic COVID-19 | 0 | 0 | 0 | 0

33. Secondary Outcome: Cohort A and Cohort B: Incidence and Severity of Symptomatic SARS-CoV-2 Infections in Seropositive Subjects During the Follow-Up Period
Time Frame: Day 30 Up to Day 225 (Approximately 8 months)
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: Placebo of R10933 + R10987 | Cohort A: R10933 + R10987 | Cohort B: Placebo of R10933 + R10987 | Cohort B: R10933 + R10987
Number analyzed (Participants) | 296 | 337 | 43 | 48
Participants
  Total Symptomatic COVID-19 | 3 | 3 | 0 | 0
  Grade 1 Symptomatic COVID-19 | 3 | 3 | 0 | 0
  Grade 2 Symptomatic COVID-19 | 0 | 0 | 0 | 0
  Grade 3Symptomatic COVID-19 | 0 | 0 | 0 | 0
  Grade 4 Symptomatic COVID-19 | 0 | 0 | 0 | 0
  Grade 5 Symptomatic COVID-19 | 0 | 0 | 0 | 0

34. Secondary Outcome: Cohort B: Number of Weeks of Symptomatic SARS-CoV-2 Infection (Broad-term) Within 14 Days of a Positive RT-qPCR at Baseline or During the EAP
Time Frame: Up to 14 Days
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | Cohort B: Placebo of R10933 + R10987 | Cohort B: R10933 + R10987
Number analyzed (Participants) | 104 | 100
weeks | 1.64 (3.493) [lower limit 3.493] | 0.90 (2.586) [lower limit 2.586]
Statistical Analysis 1: Comparison: Cohort B: Placebo of R10933 + R10987 vs Cohort B: R10933 + R10987; Test type: Superiority; p = 0.0273, Stratified Wilcoxon Rank Sum Test

35. Secondary Outcome: Cohort B: Percentage of Participants With Asymptomatic Infection Who Develop Signs and Symptoms (CDC Definition) Within 14 Days of a Positive RT-qPCR at Baseline or During the EAP
Description: as for outcome 2
Time Frame: Up to 1 month
Population: Estimate of percentage of participants meeting the criteria based on fixed categories
Measure: Number; unit: percentage of participants
Arm/Group | Cohort B: Placebo of R10933 + R10987 | Cohort B: R10933 + R10987
Number analyzed (Participants) | 104 | 100
percentage of participants | 39.7 | 26.3
Statistical Analysis 1: Comparison: Cohort B: Placebo of R10933 + R10987 vs Cohort B: R10933 + R10987; Test type: Superiority; p = 0.0460, Regression, Logistic; Odds Ratio (OR) = 0.54, 95% CI 2-sided [0.299 to 0.989]

36. Secondary Outcome: Cohort B: Percentage of Participants Who Subsequently Develop Signs and Symptoms (Strict-term) Within 14 Days of a Positive RT-qPCR at Baseline or During the EAP
Description: as for outcome 2
Time Frame: Up to 14 Days
Population: Estimate of percentage of participants meeting the criteria based on fixed categories
Measure: Number; unit: Percentage of Participants
Arm/Group | Cohort B: Placebo of R10933 + R10987 | Cohort B: R10933 + R10987
Number analyzed (Participants) | 104 | 100
Percentage of Participants | 18.5 | 9.7
Statistical Analysis 1: Comparison: Cohort B: Placebo of R10933 + R10987 vs Cohort B: R10933 + R10987; Test type: Superiority; p = 0.0721, Regression, Logistic; Odds Ratio (OR) = 0.47, 95% CI 2-sided [0.207 to 1.070]

37. Secondary Outcome: Cohort B: Number of Weeks of Symptomatic SARS-CoV-2 Infection (CDC Definition) Within 14 Days of a Positive RT-qPCR at Baseline or During the EAP
Time Frame: Up to 14 Days
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | Cohort B: Placebo of R10933 + R10987 | Cohort B: R10933 + R10987
Number analyzed (Participants) | 104 | 100
weeks | 1.71 (3.569) [lower limit 3.569] | 0.88 (2.584) [lower limit 2.584]
Statistical Analysis 1: Comparison: Cohort B: Placebo of R10933 + R10987 vs Cohort B: R10933 + R10987; Test type: Superiority; p = 0.0260, Stratified Wilcoxon Rank Sum Test

38. Secondary Outcome: Cohort B: Number of Weeks of Symptomatic SARS-CoV-2 Infection (Strict-term Definition) Within 14 Days of a Positive RT-qPCR at Baseline or During the EAP
Time Frame: Up to 14 Days
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | Cohort B: Placebo of R10933 + R10987 | Cohort B: R10933 + R10987
Number analyzed (Participants) | 104 | 100
weeks | 0.68 (1.889) [lower limit 1.889] | 0.40 (1.876) [lower limit 1.876]
Statistical Analysis 1: Comparison: Cohort B: Placebo of R10933 + R10987 vs Cohort B: R10933 + R10987; Test type: Superiority; p = 0.0614, Stratified Wilcoxon Rank Sum Test

39. Secondary Outcome: Cohort B: Change in Viral Load From Baseline to Day 8 Visit in NP Swab Samples
Time Frame: Up to day 8 visit
Measure: Least Squares Mean (Standard Error); unit: log10 copies/mL
Arm/Group | Cohort B: Placebo of R10933 + R10987 | Cohort B: R10933 + R10987
Number analyzed (Participants) | 97 | 95
log10 copies/mL | -1.543 (0.238) [lower limit 0.238] | -3.004 (0.239) [lower limit 0.239]
Statistical Analysis 1: Comparison: Cohort B: Placebo of R10933 + R10987 vs Cohort B: R10933 + R10987; Test type: Superiority; p < 0.0001, ANCOVA; LS mean difference = -1.461, 95% CI 2-sided [-2.127 to -0.795], Standard Error of Mean 0.337

40. Secondary Outcome: Cohort B: Change in Viral Load From Baseline to Day 15 Visit in NP Swab Samples
Time Frame: Up to day 15 visit
Measure: Least Squares Mean (Standard Error); unit: log10 copies/mL
Arm/Group | Cohort B: Placebo of R10933 + R10987 | Cohort B: R10933 + R10987
Number analyzed (Participants) | 97 | 95
log10 copies/mL | -4.014 (0.195) [lower limit 0.195] | -4.864 (0.199) [lower limit 0.199]
Statistical Analysis 1: Comparison: Cohort B: Placebo of R10933 + R10987 vs Cohort B: R10933 + R10987; Test type: Superiority; p = 0.0026, ANCOVA; LS mean difference = -0.850, 95% CI 2-sided [-1.400 to -0.300], Standard Error of Mean 0.279

41. Secondary Outcome: Cohort B: Time-weighted Average Change From Baseline in Viral Load (log10 Copies/mL) in NP Swab Samples Until the Day 22 Visit
Time Frame: Day 22
Measure: Least Squares Mean (Standard Error); unit: log10 copies/mL
Arm/Group | Cohort B: Placebo of R10933 + R10987 | Cohort B: R10933 + R10987
Number analyzed (Participants) | 96 | 95
log10 copies/mL | -2.639 (0.136) [lower limit 0.136] | -3.580 (0.137) [lower limit 0.137]
Statistical Analysis 1: Comparison: Cohort B: Placebo of R10933 + R10987 vs Cohort B: R10933 + R10987; Test type: Superiority; p < 0.0001, ANCOVA; LS mean difference = -0.940, 95% CI 2-sided [-1.321 to -0.559], Standard Error of Mean 0.193

42. Secondary Outcome: Cohort B: AUC in Viral Load From the First Positive SARS-CoV-2 RT-qPCR NP Swab Samples Detected During the EAP to the First Confirmed Negative Test
Time Frame: Up to 14 Days
Measure: Least Squares Mean (Standard Error); unit: log10 copies/milliLiter*days
Arm/Group | Cohort B: Placebo of R10933 + R10987 | Cohort B: R10933 + R10987
Number analyzed (Participants) | 101 | 98
log10 copies/milliLiter*days | 82.008 (4.328) [lower limit 4.328] | 55.964 (4.201) [lower limit 4.201]
Statistical Analysis 1: Comparison: Cohort B: Placebo of R10933 + R10987 vs Cohort B: R10933 + R10987; Test type: Superiority; p < 0.0001, ANCOVA; Difference of LS Mean = -26.045, 95% CI 2-sided [-37.973 to -14.117], Standard Error of Mean 6.041

43. Secondary Outcome: Cohort B: Maximum SARS-CoV-2 RT-qPCR Viral Load in NP Swab Samples in Participants With 1 or More Positive Test That Has an Onset During the EAP
Time Frame: Up to 1 month
Measure: Least Squares Mean (Standard Error); unit: log10 copies/mL
Arm/Group | Cohort B: Placebo of R10933 + R10987 | Cohort B: R10933 + R10987
Number analyzed (Participants) | 101 | 98
log10 copies/mL | 4.731 (0.238) [lower limit 0.238] | 3.336 (0.240) [lower limit 0.240]
Statistical Analysis 1: Comparison: Cohort B: Placebo of R10933 + R10987 vs Cohort B: R10933 + R10987; Test type: Superiority; p < 0.0001, ANCOVA; Difference of LS Mean = -1.395, 95% CI 2-sided [-2.063 to -0.727], Standard Error of Mean 0.338

44. Secondary Outcome: Cohort B: Number of Medically Attended Visits in Emergency Rooms or Urgent Care Centers Related to RT-qPCR Confirmed SARS-CoV-2 Infection That Has an Onset at Baseline or During the EAP
Time Frame: Up to 1 month
Measure: Mean (Standard Deviation); unit: Medically attended visits
Arm/Group | Cohort B: Placebo of R10933 + R10987 | Cohort B: R10933 + R10987
Number analyzed (Participants) | 104 | 100
Medically attended visits | 0.06 (0.234) [lower limit 0.234] | 0.00 (0.000) [lower limit 0.000]
Statistical Analysis 1: Comparison: Cohort B: Placebo of R10933 + R10987 vs Cohort B: R10933 + R10987; Test type: Superiority; p = 0.0138, Stratified Wilcoxon Rank Sum Test

45. Secondary Outcome: Cohort B: Percentage of Participants Requiring Medically Attended Visits in Emergency Rooms or Urgent Care Centers Related to a RT-qPCR Confirmed SARS CoV-2 Infection That Has an Onset at Baseline or During the EAP
Time Frame: Up to 1 month
Measure: Number; unit: Percentage of participants
Arm/Group | Cohort B: Placebo of R10933 + R10987 | Cohort B: R10933 + R10987
Number analyzed (Participants) | 104 | 100
Percentage of participants | 5.8 | 0.0
Statistical Analysis 1: Comparison: Cohort B: Placebo of R10933 + R10987 vs Cohort B: R10933 + R10987; Testing if there is an association between the observed results and treatment received; Test type: Other; p = 0.0292, Fisher Exact

46. Secondary Outcome: Cohort B: Percentage of Participants Hospitalized Related to a RT-qPCR Confirmed SARS-CoV-2 Infection That Has an Onset at Baseline or During the EAP
Time Frame: Up to 14 Days
Measure: Number; unit: Percentage of participants
Arm/Group | Cohort B: Placebo of R10933 + R10987 | Cohort B: R10933 + R10987
Number analyzed (Participants) | 104 | 100
Percentage of participants | 2.9 | 0.0
Statistical Analysis 1: Comparison: Cohort B: Placebo of R10933 + R10987 vs Cohort B: R10933 + R10987; Testing if there is an association between the observed results and treatment received; Test type: Other; p = 0.2466, Fisher Exact

47. Secondary Outcome: Cohort B: Number of Days Missed for Daily Responsibilities (Where Applicable) Due to a RT-qPCR Confirmed SARS-CoV-2 Infection That Has an Onset at Baseline or During the EAP
Time Frame: Up to 1 month
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Cohort B: Placebo of R10933 + R10987 | Cohort B: R10933 + R10987
Number analyzed (Participants) | 104 | 100
Days | 5.69 (8.802) [lower limit 8.802] | 5.18 (8.940) [lower limit 8.940]
Statistical Analysis 1: Comparison: Cohort B: Placebo of R10933 + R10987 vs Cohort B: R10933 + R10987; Test type: Superiority; p = 0.7861, Stratified Wilcoxon Rank Sum test

48. Secondary Outcome: Cohort B: Number of Days of Hospital and Intensive Care Unit (ICU) Stay in Participants Hospitalized for a RT-qPCR Confirmed SARS-CoV-2 Infection That Has an Onset at Baseline or During the EAP
Time Frame: Up to 1 month
Population: Estimate of proportion of participants meeting the criteria
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Cohort B: Placebo of R10933 + R10987 | Cohort B: R10933 + R10987
Number analyzed (Participants) | 104 | 100
days | 0.38 (2.671) [lower limit 2.671] | 0.00 (0.000) [lower limit 0.000]
Statistical Analysis 1: Comparison: Cohort B: Placebo of R10933 + R10987 vs Cohort B: R10933 + R10987; Test type: Superiority; p = 0.0842, Stratified Wilcoxon Rank Sum test

49. Secondary Outcome: Concentrations of REGN10987 in Serum Over Time (Cohort A)
Time Frame: 0 Days Post-Dose, 28 Days Post-Dose, 56 Days Post-Dose, 112 Days Post-Dose
Population: Number of participants in Cohort A with reportable concentrations obtained from baseline to day 112 of study for REGN10987 only. This PK analysis set (PKAS: Safety Subset) includes all treated subjects who received any study drug and had at least 1 non-missing imdevimab measurement following study drug administration. The PK analysis safety subset is based on the actual treatment received (as treated) rather than as randomized
Measure: Mean (Standard Deviation); unit: milligrams per Liter (mg/L)
Arm/Group | Cohort A: R10933 + R10987
Number analyzed (Participants) | 138
milligrams per Liter (mg/L)
  0 Days Post-Dose (n=107): number analyzed (Participants) | 107
  0 Days Post-Dose (n=107) | 0.0233 (0.145)
  28 Days Post-Dose (n=74): number analyzed (Participants) | 74
  28 Days Post-Dose (n=74) | 24.6 (9.78)
  56 Days Post-Dose (n=105): number analyzed (Participants) | 105
  56 Days Post-Dose (n=105) | 10.4 (5.88)
  112 Days Post-Dose (n=88): number analyzed (Participants) | 88
  112 Days Post-Dose (n=88) | 2.10 (1.68)

50. Secondary Outcome: Concentrations of REGN10987 in Serum Over Time (Cohort B)
Time Frame: 0 Days Post-Dose, 28 Days Post-Dose, 56 Days Post-Dose, 112 Days Post-Dose
Population: Number of participants in Cohort B with reportable concentrations obtained from baseline to day 112 of study for REGN10987 only. This PK analysis set (PKAS: Safety Subset) includes all treated subjects who received any study drug and had at least 1 non-missing imdevimab measurement following study drug administration. The PK analysis safety subset is based on the actual treatment received (as treated) rather than as randomized
Measure: Mean (Standard Deviation); unit: milligrams per Liter (mg/L)
Groups:
- Cohort B: R10933 + R10987: Cohort B: R10933 + R10987 Adult and Adolescent Participants (≥12years) Who Are SARS-CoV-2 RT-qPCR negative at baseline
Arm/Group | Cohort B: R10933 + R10987
Number analyzed (Participants) | 9
milligrams per Liter (mg/L)
  0 Days Post-Dose (n=7): number analyzed (Participants) | 7
  0 Days Post-Dose (n=7) | 0 (0)
  28 Days Post-Dose (n=6): number analyzed (Participants) | 6
  28 Days Post-Dose (n=6) | 31.0 (8.26)
  56 Days Post-Dose (n=8): number analyzed (Participants) | 8
  56 Days Post-Dose (n=8) | 14.0 (6.20)
  112 Days Post-Dose (n=5): number analyzed (Participants) | 5
  112 Days Post-Dose (n=5) | 4.62 (3.30)

51. Secondary Outcome: Concentrations of REGN10933 in Serum Over Time (Cohort A)
Time Frame: 0 Days Post-Dose, 28 Days Post-Dose, 56 Days Post-Dose, 112 Days Post-Dose
Population: Number of participants in Cohort A with reportable concentrations obtained from baseline to day 112 of study for REGN10933 only. This PK analysis set (PKAS: Safety Subset) includes all treated subjects who received any study drug and had at least 1 non-missing imdevimab measurement following study drug administration. The PK analysis safety subset is based on the actual treatment received (as treated) rather than as randomized
Measure: Mean (Standard Deviation); unit: milligrams per Liter (mg/L)
Arm/Group | Cohort A: R10933 + R10987
Number analyzed (Participants) | 138
milligrams per Liter (mg/L)
  0 Days Post-Dose (n=107): number analyzed (Participants) | 107
  0 Days Post-Dose (n=107) | 0.0190 (0.123)
  28 Days Post-Dose (n=73): number analyzed (Participants) | 73
  28 Days Post-Dose (n=73) | 30.8 (12.0)
  56 Days Post-Dose (n=106): number analyzed (Participants) | 106
  56 Days Post-Dose (n=106) | 14.8 (7.18)
  112 Days Post-Dose (n=88): number analyzed (Participants) | 88
  112 Days Post-Dose (n=88) | 3.61 (2.46)

52. Secondary Outcome: Concentrations of REGN10933 in Serum Over Time (Cohort B)
Time Frame: 0 Days Post-Dose, 28 Days Post-Dose, 56 Days Post-Dose, 112 Days Post-Dose
Population: Number of participants in Cohort B with reportable concentrations obtained from baseline to day 112 of study for REGN10933 only. This PK analysis set (PKAS: Safety Subset) includes all treated subjects who received any study drug and had at least 1 non-missing imdevimab measurement following study drug administration. The PK analysis safety subset is based on the actual treatment received (as treated) rather than as randomized
Measure: Mean (Standard Deviation); unit: milligrams per Liter (mg/L)
Arm/Group | Cohort B: R10933 + R10987
Number analyzed (Participants) | 9
milligrams per Liter (mg/L)
  0 Days Post-Dose (n=7): number analyzed (Participants) | 7
  0 Days Post-Dose (n=7) | 0 (0)
  28 Days Post-Dose (n=6): number analyzed (Participants) | 6
  28 Days Post-Dose (n=6) | 37.6 (13.3)
  56 Days Post-Dose (n=8): number analyzed (Participants) | 8
  56 Days Post-Dose (n=8) | 19.1 (9.50)
  112 Days Post-Dose (n=3): number analyzed (Participants) | 3
  112 Days Post-Dose (n=3) | 4.58 (3.02)

53. Secondary Outcome: Immunogenicity as Measured by Anti-drug Antibodies (ADAs) to REGN10933
Time Frame: Up to 8 months
Population: This ADA analysis set (AAS) includes all treated subjects who received study drug and had at least 1 non-missing ADA result after study drug administration. The AAS is based on the actual treatment received.
Measure: Count of Participants; unit: Participants
Groups:
- Placebo: Overall Adult and Adolescent Subjects (≥12years) Who Are SARS-CoV-2 RT-qPCR negative at baseline
- R10933 + R10987: Participants received a single 1200mg intravenous dose of REGN10933+REGN10987
Arm/Group | Placebo | R10933 + R10987
Number analyzed (Participants) | 1606 | 1595
Participants | 1544 | 1319

54. Secondary Outcome: Immunogenicity as Measured by Anti-drug Antibodies (ADAs) to REGN10987
Time Frame: Up to 8 months
Population: as for outcome 53
Measure: Count of Participants; unit: Participants
Groups:
- R10987 +R10933: Participants received a single 1200mg intravenous dose of REGN10933+REGN10987
Arm/Group | Placebo | R10987 +R10933
Number analyzed (Participants) | 1606 | 1595
Participants | 1500 | 1251

55. Secondary Outcome: Immunogenicity as Measured by Neutralizing Anti-drug Antibody (NAb) to REGN10933
Description: (TE&TB+;NAb+) = TE = Treatment-Emergent; TB = Treatment-boosted; NAb+ = Positive in NAb assay
Time Frame: Up to 8 months
Population: This ADA analysis set (AAS) includes all treated participants who received study drug and had at least 1 non-missing ADA result after study drug administration. The AAS is based on the actual treatment received.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | R10933 + R10987
Number analyzed (Participants) | 1606 | 1595
Participants | 4 | 33

56. Secondary Outcome: Immunogenicity as Measured by Neutralizing Anti-drug Antibody (NAb) to REGN10987
Description: (TE&TB+;NAb+) = TE = Treatment-emergent; TB = Treatment-boosted; NAb+ = Positive in NAb assay
Time Frame: Up to 8 Months
Population: as for outcome 53
Measure: Count of Participants; unit: Participants
Groups:
- R10987 + R10987: Participants received a single 1200mg intravenous dose of REGN10933+REGN10987
Arm/Group | Placebo | R10987 + R10987
Number analyzed (Participants) | 1606 | 1595
Participants | 27 | 160

ADVERSE EVENTS:
Time Frame: Up to day 226
Groups:
- Cohort A Placebo: Cohort A: Placebo of R10933 + R10987 Adult and Adolescent Subjects (≥12years) Who Are SARS-CoV-2 RT-qPCR negative at baseline
- Cohort A R10933+R10987: Cohort A: R10933 + R10987 Adult and Adolescent Subjects (≥12years) Who Are SARS-CoV-2 RT-qPCR negative at baseline
- Cohort A1 Placebo: Cohort A1: Placebo of R10933 + R10987 Pediatric Subjects (<12 years) with SARS-CoV-2 RT-qPCR Negative
- Cohort B Placebo: Cohort B: Placebo of R10933 + R10987 Adult and Adolescent Subjects (≥12years) Who Are SARS-CoV-2 RT-qPCR Positive
- Cohort B R10933+R10987: Cohort B: R10933 + R10987 Adult and Adolescent Subjects (≥12years) who Are SARS-CoV-2 RT-qPCR Positive
- Undetermined Placebo: Undetermined: Placebo of R10933 + R10987 Adult and Adolescent subjects (≥12 years) whose baseline RT-qPCR status was inconclusive or missing
- Undetermined R10933+R10987: Undetermined: R10933 + R10987 Adult and Adolescent subjects (≥12 years) whose baseline RT-qPCR status was inconclusive or missing
Arm/Group | Cohort A Placebo | Cohort A R10933+R10987 | Cohort A1 Placebo | Cohort B Placebo | Cohort B R10933+R10987 | Undetermined Placebo | Undetermined R10933+R10987
All-Cause Mortality (participants affected / at risk) | 2/1428 | 3/1439 | 0/1 | 0/170 | 0/165 | 0/44 | 0/23
Serious Adverse Events (participants affected / at risk) | 23/1428 | 24/1439 | 0/1 | 5/170 | 1/165 | 0/44 | 0/23
Other Adverse Events (participants affected / at risk) | 247/1428 | 96/1439 | 0/1 | 63/170 | 41/165 | 10/44 | 2/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A Placebo (N=1428) | Cohort A R10933+R10987 (N=1439) | Cohort A1 Placebo (N=1) | Cohort B Placebo (N=170) | Cohort B R10933+R10987 (N=165) | Undetermined Placebo (N=44) | Undetermined R10933+R10987 (N=23)
COVID-19 (Infections and infestations) | 5 (5) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Scrotal abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abscess limb (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gangrene (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Soft tissue infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gun shot wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Soft tissue injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Burns second degree (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post procedural inflammation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Traumatic lung injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mania (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Schizophrenia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Essential hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertensive urgency (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cervix carcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast haematoma (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A Placebo (N=1428) | Cohort A R10933+R10987 (N=1439) | Cohort A1 Placebo (N=1) | Cohort B Placebo (N=170) | Cohort B R10933+R10987 (N=165) | Undetermined Placebo (N=44) | Undetermined R10933+R10987 (N=23)
COVID-19 (Infections and infestations) | 148 (149) | 29 (32) | 0 (0) | 58 (59) | 35 (35) | 4 (4) | 1 (1)
Asymptomatic COVID-19 (Infections and infestations) | 119 (119) | 71 (73) | 0 (0) | 6 (6) | 7 (7) | 7 (7) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator has the right to independently publish study results from the investigator's site after a multi-center publication, or a defined period after the completion of the study by all sites. The investigator must provide the sponsor a copy of any such publication derived from the study for review and comment in advance of any submission, and delay publication, if requested, to allow the Sponsor to preserve its proprietary rights.

DOCUMENTS (3):
  • Study Protocol (2021-03-25): https://cdn.clinicaltrials.gov/large-docs/18/NCT04452318/Prot_001.pdf
  • Statistical Analysis Plan (2021-03-26): https://cdn.clinicaltrials.gov/large-docs/18/NCT04452318/SAP_002.pdf
  • Informed Consent Form (2021-01-22): https://cdn.clinicaltrials.gov/large-docs/18/NCT04452318/ICF_000.pdf